CLINICAL TRIAL: NCT04117620
Title: Validity of the French Version of the Child's Vestibular Disorder Symptoms Questionnaire
Acronym: QEV-FR
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP190616; ID RCB : 2019-A00364-53 (Other: ANSM)
Record Dates: First submitted 2019-10-03; First posted 2019-10-07 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Dizziness
Keywords: Pediatric vestibular symptom; Pediatric vestibular symptom questionnaire in french
MeSH Terms: conditions — Dizziness | interventions — Patient Health Questionnaire

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients: Patients from 7 to 17 years of age with vestibular deficiency.
  Interventions: Other: Pediatric Vestibular Symptom Questionnaire
- Controls: Subjects from 7 to 17 years of age without vestibular deficiency
  Interventions: Other: Pediatric Vestibular Symptom Questionnaire

INTERVENTIONS:
Other: Pediatric Vestibular Symptom Questionnaire — Subjects respond to the translated questionnaire twice with 15 days interval
  Other Names: Patient questionnaire

SUMMARY:
There is currently no score in French for evaluating disorders of the child's balance. Only one questionnaire was validated in the child in English in 2016, the " Pediatric Vestibular Symptom Questionnaire ". The objective of the research is to validate the French translation of this questionnaire.

DETAILED DESCRIPTION:
Balance disorders are the most common cause of dizziness in children with a prevalence of 0.7 to 15%. Vestibular migraine, benign paroxysmal positional vertigo of the child, post-concussion dizziness as a result of cranial trauma, and viral vestibular neuritis are the most common causes. However, these disorders are often undiagnosed in children as many doctors may attribute these symptoms to behavioural disorders or clumsiness. This is probably because of the difficulty children may have in expressing or describing their dizziness symptoms without specific questioning, but also because of the tendency of children to accept the terminology that an adult offers them or even tend to cling to their parents when they experience a balance disorder or vertigo. Vestibular disorders can also have secondary psychological symptoms with an impact on school learning and quality of life. A precise interrogation to check the symptoms, to look for the triggers and to trace the installation of the symptoms is fundamental to diagnose and make a therapeutic decision. Thus, it is very important to help the child express his or her feelings by proposing different descriptions and formulations to determine the etiology and diagnosis. While a number of international questionnaires validated and translated into French exist in the adult to assess the presence, severity and impact of vestibular symptoms, there is currently no score in French for evaluating disorders of the child's balance. Only one questionnaire was validated in the child in English in 2016, the " Pediatric Vestibular Symptom Questionnaire ". The objective of the research is to validate the French translation of this questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Non-opposition of the holders of parental authority and the subject to participation in the study
* Subjects between 7 and 17 years of age
* Patients : patients followed in the clinic at Necker Hospital in pediatric department of otolaryngology and cervico-facial surgery and presenting with dizziness without associated ophthalmological or neurological disorder.
* Controls : subject with no vestibular deficiency, symptoms of balance disorder, migraine, otological pathology or ophthalmological disorder at the time of inclusion or background.

Exclusion Criteria:

- Absence of diagnosis after etiological assessment.

Ages: 7 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients followed by the department of otolaryngology and cervico-facial surgery of Necker-Enfants Malades hospital and siblings for the control subjects.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2021-04-28 (Actual); Study Completion 2021-04-28 (Actual)

PRIMARY OUTCOMES:
Reproducibility | 1 year
  Reproducibility of the questionnaire completed by a subject at 15 days apart. Student t-test.
Consistency reliability test | 1 year
  Measure of efficiency. Comparison of questionnaires completed by patients and controls.
Item-total Pearson correlation | 1 year
  Measure of efficiency. Comparison of questionnaires completed by patients and controls.
Principal components analysis | 1 year
  Measure of efficiency. Comparison of questionnaires completed by patients and controls.

CONTACTS AND LOCATIONS:
Overall Officials: François Simon, MD MSc, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP, Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rigal T, Parodi M, Brisse F, Denoyelle F, Loundon N, Simon F. Translation and validation of the PVSQ and DHI-PC questionnaires for pediatric dizziness. Eur Ann Otorhinolaryngol Head Neck Dis. 2024 Jan;141(1):5-12. doi: 10.1016/j.anorl.2023.05.001. Epub 2023 May 22. PMID 37225531